CLINICAL TRIAL: NCT02575807
Title: A Phase 1/2, Open-Label Safety and Efficacy Evaluation of CRS-207 in Combination With Epacadostat in Adults With Platinum-Resistant Ovarian, Fallopian, or Peritoneal Cancer
Brief Title: Safety and Efficacy of CRS-207 With Epacadostat in Platinum Resistant Ovarian, Fallopian or Peritoneal Cancer
Acronym: SEASCAPE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was stopped due to low enrollment and lack of clinical activity.
Sponsor: Aduro Biotech, Inc. (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADU-CL-11
Record Dates: First submitted 2015-10-12; First posted 2015-10-15 (Estimated); Results first posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Platinum-resistant Ovarian Cancer; Platinum-resistant Fallopian Cancer; Platinum-resistant Peritoneal Cancer
Keywords: Ovarian cancer; Fallopian cancer; Primary peritoneal cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — epacadostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1: CRS-207 (Experimental): CRS-207 administered in 3-week cycles.
  * CRS-207 (1 x 10e9 colony forming units [CFU]) administered by intravenous (IV) infusion. For Cycle 1 through Cycle 6, CRS-207 will be administered on Day 1 of each cycle. After 6 cycles, CRS-207 will be administered on Day 1 once every 6 weeks (every other cycle).
  Interventions: Biological: CRS-207
- Phase 1: CRS-207/IDO 100 mg (Experimental): CRS-207 administered in 3-week cycles, IDO administered twice daily (BID).
  * CRS-207 (1 x 10e9 CFU) administered by IV infusion. For Cycle 1 through Cycle 6, CRS-207 administered on Day 1 of each cycle. After 6 cycles, CRS-207 administered on Day 1 once every 6 weeks (every other cycle).
  * IDO (100 milligrams [mg]) administered by mouth (PO) BID, starting on Day 2 of the first CRS-207 treatment cycle.
  Interventions: Biological: CRS-207; Drug: Epacadostat
- Phase 1: CRS-207/IDO 300 mg (Experimental): CRS-207 administered in 3-week cycles, IDO administered BID.
  * CRS-207 (1 x 10e9 CFU) administered by IV infusion. For Cycle 1 through Cycle 6, CRS-207 administered on Day 1 of each cycle. After 6 cycles, CRS-207 administered on Day 1 once every 6 weeks (every other cycle).
  * IDO (300 mg) administered PO BID, starting on Day 2 of the first CRS-207 treatment cycle.
  Interventions: Biological: CRS-207; Drug: Epacadostat
- Phase 2: CRS-207/Pembro/IDO (Experimental): CRS-207 and pembrolizumab (pembro) administered in 3-week cycles, IDO administered BID.
  * CRS-207 (1 x 10e9 CFU) administered by IV infusion. For Cycle 1 through Cycle 6, CRS-207 administered on Day 2 of each cycle. After 6 cycles, CRS-207 administered on Day 2 once every 6 weeks (every other cycle).
  * Pembro (200 mg) administered by IV infusion on Day 1 in 3-week cycles.
  * IDO (300 mg) administered PO BID, starting on Day 3 of the first CRS-207 treatment cycle.
  Interventions: Biological: CRS-207; Drug: Epacadostat; Biological: Pembrolizumab
- Phase 2: CRS-207/Pembro (Experimental): CRS-207 and pembro administered in 3-week cycles.
  * CRS-207 (1 x 10e9 CFU) administered by IV infusion. For Cycle 1 through Cycle 6, CRS-207 administered on Day 2 of each cycle. After 6 cycles, CRS-207 administered on Day 2 once every 6 weeks (every other cycle).
  * Pembro (200 mg) administered by IV infusion on Day 1 in 3-week cycles.
  Interventions: Biological: CRS-207; Biological: Pembrolizumab

INTERVENTIONS:
Biological: CRS-207 — via IV infusion
  Other Names: Live, attenuated double-deleted Listeria monocytogenes (LADD)
Drug: Epacadostat — PO BID
  Other Names: INCB024360; IDO
  Arms: Phase 1: CRS-207/IDO 100 mg; Phase 1: CRS-207/IDO 300 mg; Phase 2: CRS-207/Pembro/IDO
Biological: Pembrolizumab — via IV infusion
  Other Names: Keytruda®; Pembro
  Arms: Phase 2: CRS-207/Pembro; Phase 2: CRS-207/Pembro/IDO

SUMMARY:
This 2-part, Phase 1/2 study will test investigational cancer drugs known as CRS-207, epacadostat (IDO), and pembrolizumab (pembro). The purpose of this study is to find out how safe it is to give the investigational drugs to women with platinum-resistant ovarian, fallopian tube, or peritoneal cancer and if it helps patients with these types of cancer live longer or can help shrink or slow the growth of cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed disease

   * Phase 1: Individuals with epithelial ovarian cancer, fallopian tube carcinoma, or primary peritoneal carcinomas who are considered to have platinum-resistant disease (progression within 6 months from completion of platinum-based chemotherapy).
   * Phase 2: Individuals with epithelial ovarian cancer, fallopian tube carcinoma, or primary peritoneal carcinomas who are considered to have platinum-resistant disease (progression within 6 months from completion of a minimum of 4 platinum therapy cycles).
2. Measurable disease, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
3. Agree to provide core biopsies at baseline and at Cycle 2 Day 15
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Available archived tumor tissue for central analysis
6. Adequate organ and marrow function

Exclusion Criteria

1. Platinum-refractory disease (progression during the first platinum-based chemotherapy)
2. Major surgical procedure within 4 weeks prior to Study Day 1
3. Inaccessible tumors or for whom biopsy is contraindicated
4. Clinically significant ascites
5. Phase 2 only: Previous treatment with >3 chemotherapy regimens for locally advanced or metastatic disease
6. Active bowel obstruction, or hospitalization for bowel obstruction within 2 months prior to screening
7. Require parenteral nutrition
8. Hospitalization within 2 weeks prior to screening
9. Received any anticancer medication or therapy in the 21 days prior to study Day 1
10. Prior monoclonal antibody treatment within 4 weeks before study Day 1
11. History of listeriosis or previous treatment with a listeria-based immunotherapy
12. Known allergy to both penicillin and sulfa antibiotics
13. Any immunodeficiency disease or immune-compromised state
14. Received prior immune checkpoint inhibitors (e.g., anti-CTLA-4, anti-PD-1, anti PDL-1) and any other antibody or drug specifically targeting T-cell costimulation or an IDO inhibitor
15. Pregnant or breastfeeding
16. Clinically significant heart disease
17. Valvular heart disease that requires antibiotic prophylaxis for prevention of endocarditis
18. History of any autoimmune disease which required systemic therapy in the past 2 years
19. Diagnosed with another malignancy within the past 3 years
20. Currently receiving therapy with a UDP-glucuronosyltransferase 1A9 inhibitor including diclofenac, imipramine, ketoconazole, mefenamic acid, and probenecid
21. Receiving monoamine oxidase inhibitor (MAOIs) or a drug which has significant MAOI activity (meperidine, linezolid, methylene blue) within the 21 days before screening
22. Had prior serotonin syndrome
23. Has implanted medical devices that pose high risks for colonization and cannot be easily removed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (10):
  - Scottsdale Healthcare Hospitals DBA HonorHealth, Scottsdale, Arizona
  - Stanford Cancer Center, Stanford, California
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHUM - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: CRS-207/IDO 100 mg: CRS-207 administered in 3-week cycles, epacadostat (IDO) administered twice daily (BID).
  * CRS-207 (1 x 10e9 CFU) administered by IV infusion. For Cycle 1 through Cycle 6, CRS-207 administered on Day 1 of each cycle. After 6 cycles, CRS-207 administered on Day 1 once every 6 weeks (every other cycle).
  * IDO (100 milligrams [mg]) administered by mouth (PO) BID, starting on Day 2 of the first CRS-207 treatment cycle.
Period: Overall Study
Arm/Group | Phase 1: CRS-207 | Phase 1: CRS-207/IDO 100 mg | Phase 1: CRS-207/IDO 300 mg | Phase 2: CRS-207/Pembro/IDO | Phase 2: CRS-207/Pembro
Started | 9 | 4 | 16 | 2 | 4
Treated (Subjects who received at least 1 dose of protocol-specified drug.) | 8 | 4 | 16 | 1 | 3
Completed (No predetermined study completion date or study completion event specified in protocol.) | 0 (Subjects followed until lost to follow-up/consent withdrawn/study termination/death.) | 0 (Subjects followed until lost to follow-up/consent withdrawn/study termination/death.) | 0 (Subjects followed until lost to follow-up/consent withdrawn/study termination/death.) | 0 (Subjects followed until lost to follow-up/consent withdrawn/study termination/death.) | 0 (Subjects followed until lost to follow-up/consent withdrawn/study termination/death.)
Not Completed | 9 | 4 | 16 | 2 | 4
Not completed — Death | 8 | 3 | 7 | 0 | 1
Not completed — Study terminated by Sponsor | 0 | 1 | 7 | 0 | 1
Not completed — Terminated due to FDA clinical hold | 1 | 0 | 0 | 0 | 0
Not completed — Terminated due to physician decision | 0 | 0 | 1 | 0 | 0
Not completed — Subject ineligible - medical implant | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis provided for all subjects who were administered at least 1 dose of protocol-specified drug (the Safety Analysis Set [SAF]).
Groups:
- Phase 1: CRS-207: CRS-207 administered in 3-week cycles.
  * CRS-207 (1 x 10e9 CFU) administered by IV infusion. For Cycle 1 through Cycle 6, CRS-207 will be administered on Day 1 of each cycle. After 6 cycles, CRS-207 will be administered on Day 1 once every 6 weeks (every other cycle).
- Phase 1: CRS-207/IDO 100 mg: CRS-207 administered in 3-week cycles, IDO administered BID.
  * CRS-207 (1 x 10e9 CFU) administered by IV infusion. For Cycle 1 through Cycle 6, CRS-207 administered on Day 1 of each cycle. After 6 cycles, CRS-207 administered on Day 1 once every 6 weeks (every other cycle).
  * IDO (100 mg) administered PO BID, starting on Day 2 of the first CRS-207 treatment cycle.
- Phase 2: CRS-207/Pembro/IDO: CRS-207 and pembro administered in 3-week cycles, IDO administered BID.
  * CRS-207 (1 x 10e9 CFU) administered by IV infusion. For Cycle 1 through Cycle 6, CRS-207 administered on Day 2 of each cycle. After 6 cycles, CRS-207 administered on Day 2 once every 6 weeks (every other cycle).
  * Pembro (200 mg) administered by IV infusion on Day 1 in 3-week cycles.
  * IDO (300 mg) administered PO BID, starting on Day 3 of the first CRS-207 treatment cycle.
- Total: Total of all reporting groups
Arm/Group | Phase 1: CRS-207 | Phase 1: CRS-207/IDO 100 mg | Phase 1: CRS-207/IDO 300 mg | Phase 2: CRS-207/Pembro/IDO | Phase 2: CRS-207/Pembro | Total
Number analyzed (Participants) | 8 | 4 | 16 | 1 | 3 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (11.03) | 62.0 (12.99) | 62.4 (9.35) | 60.0 (NA) — Only 1 subject in the SAF for this study arm; standard deviation could not be calculated | 61.7 (5.13) | 61.9 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 16 | 1 | 3 | 32
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 7 | 4 | 15 | 1 | 3 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 8 | 3 | 15 | 1 | 2 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 0 | 2 | 0 | 0 | 2
  United States | 8 | 4 | 14 | 1 | 3 | 30

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Subjects Reporting Hematologic and/or Non-hematologic Dose-limiting Toxicity (DLT)
Description: Count of subjects in the Phase 1 cohorts who reported a hematologic and/or non-hematologic DLT. Non-hematological DLTs are defined as follows, excluding the safety events specified for exemption in Section 5.3.1 of the study protocol:
  * any treatment-emergent adverse event (TEAE) not attributable to disease or disease-related processes that occurs during the DLT observation period (Cycle 1) and is Grade 3 or higher according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4;
  * any use of systemic steroids; and/or
  * a study drug dose interruption lasting ≥ 7 days for an adverse event with an unclear relationship to study drug.
  Hematological DLTs are defined as:
  * Grade 4 neutropenia lasting >7 days;
  * Grade ≥3 febrile neutropenia;
  * Grade 4 anemia;
  * Grade 4 thrombocytopenia or ≥ Grade 3 thrombocytopenia lasting >7 days or associated with bleeding; and/or
  * Dose delay >7 days secondary to myelosuppression.
Time Frame: Subjects followed for DLTs for 21 days following the first dose of CRS-207 (treatment Cycle 1 for CRS-207).
Population: Analysis performed on subjects in the Phase 1 safety analysis set (SAF).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: CRS-207 | Phase 1: CRS-207/IDO 100 mg | Phase 1: CRS-207/IDO 300 mg
Number analyzed (Participants) | 8 | 4 | 16
Participants | 1 | 0 | 1

2. Primary Outcome: Phase 1: Adverse Events (AEs) by CTCAE Grade 3 or Higher
Description: Count of subjects in the Phase 1 cohorts with incidences of CTCAE Grade 3 or higher AEs.
Time Frame: Subjects followed from the start of study treatment until 30 days following the final dose of study drug, an average of 3 months.
Population: Analysis performed on subjects in the Phase 1 safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: CRS-207 | Phase 1: CRS-207/IDO 100 mg | Phase 1: CRS-207/IDO 300 mg
Number analyzed (Participants) | 8 | 4 | 16
Participants | 6 | 3 | 14

3. Primary Outcome: Phase 2: Adverse Events (AEs)
Description: Count of subjects in the Phase 2 cohorts with incidences of AEs.
Time Frame: Subjects followed from the start of study treatment until 30 days following the final dose of study drug, an average of 2 months.
Population: Analysis performed on subjects in the Phase 2 safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: CRS-207/Pembro/IDO | Phase 2: CRS-207/Pembro
Number analyzed (Participants) | 1 | 3
Participants | 1 | 3

4. Primary Outcome: Phase 2: Objective Response Rate (ORR)
Description: ORR was evaluated for Phase 2 subjects based upon the best overall response (BOR) for individual study subjects. BOR was determined by the highest post-baseline qualitative response value for each assessed subject as measured by modified response evaluation criteria in solid tumors (mRECIST) and given the following hierarchy of overall response results: complete response (CR) > partial response (PR) > stable disease (SD) > progressive disease (PD) > not evaluable (NE). The protocol-specified ORR was defined as the percentage of evaluable subjects with a BOR of CR or PR; however, this percentage was not calculated per the final study Statistical Analysis Plan (SAP). Therefore, the number of evaluable subjects with BOR mRECIST values of CR, PR, SD, PD, and NE are provided for this outcome measure.
Time Frame: BOR was assessed from the first dose of study treatment until documented disease progression, initiation of a new cancer treatment, death, or study termination, whichever comes first, assessed up to 20 weeks.
Population: Analysis performed on subjects in the SAF who had ≥1 post-baseline response assessment. One subject in the Phase 2 SAF did not complete ≥1 post-baseline response assessment and was therefore not evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: CRS-207/Pembro/IDO | Phase 2: CRS-207/Pembro
Number analyzed (Participants) | 1 | 2
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0
  Stable Disease | 0 | 0
  Progressive Disease | 1 | 2
  Not Evaluable | 0 | 0

5. Secondary Outcome: Phase 1: Objective Response Rate (ORR) by mRECIST
Description: ORR was evaluated for Phase 1 subjects based upon the best overall response (BOR) for individual study subjects. BOR was determined by the highest post-baseline qualitative response value for each assessed subject as measured by modified response evaluation criteria in solid tumors (mRECIST), RECIST v1.1, and GCIG CA-125 criteria and given the following hierarchy of overall response results: complete response (CR) > partial response (PR) > stable disease (SD) > progressive disease (PD) > not evaluable (NE). The protocol-specified ORR was defined as the percentage of evaluable subjects with a BOR of CR or PR; however, this percentage was not calculated per the final study Statistical Analysis Plan (SAP). Therefore, the number of evaluable subjects with BOR mRECIST values of CR, PR, SD, PD, and NE are provided for this outcome measure.
Time Frame: BOR was assessed from the first dose of study treatment until documented disease progression, starting of a new cancer treatment, death, or study termination, whichever is earlier, assessed up to 100 weeks.
Population: Analysis performed on subjects in the SAF who had ≥1 post-baseline response assessment. Three subjects in the Phase 1 SAF did not complete ≥1 post-baseline response assessment and were therefore not evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: CRS-207 | Phase 1: CRS-207/IDO 100 mg | Phase 1: CRS-207/IDO 300 mg
Number analyzed (Participants) | 8 | 4 | 13
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0
  Stable Disease | 1 | 1 | 4
  Progressive Disease | 7 | 3 | 6
  Not Evaluable | 0 | 0 | 3

6. Secondary Outcome: Phase 1: Progression Free Survival (PFS)
Description: Number of weeks from the date of first dose of study treatment to the first date of objectively determined progressive disease (PD) or death due to any cause, estimated using Kaplan-Meier (KM) methods with 95% confidence intervals (CIs). PD is determined by mRECIST, RECIST v1.1, and GCIG CA-125.
Time Frame: Subjects followed for disease progression from first dose of study treatment until 30 days after last dose of study treatment or initiation of new cancer treatment, whichever comes first, assessed up to 100 weeks
Population: Analysis performed on subjects in the Phase 1 SAF.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 1: CRS-207 | Phase 1: CRS-207/IDO 100 mg | Phase 1: CRS-207/IDO 300 mg
Number analyzed (Participants) | 8 | 4 | 16
weeks | 8.43 [3.00 to 9.71] | 4.71 [3.29 to 17.14] | 8.43 [4.29 to 36.00]

7. Secondary Outcome: Disease Control Rate (DCR)
Description: The protocol-specified DCR was defined as the percentage of evaluable subjects with a BOR of CR or PR, or SD as determined by mRECIST, RECIST v1.1, and GCIG CA-125 criteria.
Time Frame: BOR was assessed from the first dose of study treatment until documented disease progression, starting of a new cancer treatment, death, or study termination, whichever comes first, assessed up to 100 weeks.
Population: Analysis performed on subjects in the Phase 1 and Phase 2 SAF.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: CRS-207 | Phase 1: CRS-207/IDO 100 mg | Phase 1: CRS-207/IDO 300 mg | Phase 2: CRS-207/Pembro/IDO | Phase 2: CRS-207/Pembro
Number analyzed (Participants) | 8 | 4 | 16 | 1 | 3
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0 | 0
  Stable Disease (SD) | 1 | 1 | 4 | 0 | 0

8. Secondary Outcome: Duration of Response (DOR)
Description: Number of weeks from date of CR or PR designation until PD designation, as determined by mRECIST, RECIST v1.1 and GCIG CA-125 criteria.
Time Frame: Subjects followed for disease progression from date of CR or PR designation until documented disease progression or study termination, whichever comes first, assessed up to 100 weeks.
Population: No study subjects achieved CR or PR designation; therefore, per the final SAP DOR was not derived.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: CRS-207 | Phase 1: CRS-207/IDO 100 mg | Phase 1: CRS-207/IDO 300 mg | Phase 2: CRS-207/Pembro/IDO | Phase 2: CRS-207/Pembro
Number analyzed (Participants) | 8 | 4 | 16 | 1 | 3
Participants | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Overall Survival (OS)
Description: Number of weeks from the date of first dose of study treatment to the date of death from any cause, estimated using KM methods with 95% CIs for subjects in the SAF. Subjects without documentation of death at the time of analysis were censored as of the date the subject was last known to be alive. For subjects lost to follow up, the last visit or last contact date where the subject is documented to be alive will be used to estimate last known date alive.
Time Frame: OS was assessed from the first dose of study treatment until death or study termination, whichever comes first, assessed up to 100 weeks.
Population: Analysis performed on subjects in the Phase 1 and Phase 2 SAF.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 1: CRS-207 | Phase 1: CRS-207/IDO 100 mg | Phase 1: CRS-207/IDO 300 mg | Phase 2: CRS-207/Pembro/IDO | Phase 2: CRS-207/Pembro
Number analyzed (Participants) | 8 | 4 | 16 | 1 | 3
weeks | 49.07 [4.71 to 69.29] | 30.00 [18.71 to 88.71] | 27.00 [18.14 to 51.29] | 9.29 | 18.43 [10.43 to 18.57]

10. Primary Outcome: Phase 2: Progression Free Survival (PFS)
Description: Number of weeks from the date of first dose of study treatment to the first date of objectively determined progressive disease (PD) or death from any cause, estimated using Kaplan-Meier (KM) methods with 95% confidence intervals (CIs). PD is determined by mRECIST.
Time Frame: Subjects followed for disease progression from first dose of study treatment until 30 days after last dose of study treatment or initiation of new cancer treatment, whichever comes first, assessed up to 20 weeks.
Population: Analysis performed on subjects in the Phase 2 SAF.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: CRS-207/Pembro/IDO | Phase 2: CRS-207/Pembro
Number analyzed (Participants) | 1 | 3
weeks | 5.71 | 7.36 [6.14 to 8.57]

ADVERSE EVENTS:
Time Frame: Subjects were followed for serious and non-serious adverse events (AEs) from the beginning of any study drug until 30 days following the last dose of study drug, an average of 3 months. Subjects were followed for survival until withdrawal of consent, loss to follow-up, death, or study termination (whichever is first), an average of 35 weeks.
Description: AEs reported for the Safety Analysis Set (SAF). Methods of determining whether certain AEs have occurred include regular investigator assessment and regular laboratory testing.
Arm/Group | Phase 1: CRS-207 | Phase 1: CRS-207/IDO 100 mg | Phase 1: CRS-207/IDO 300 mg | Phase 2: CRS-207/Pembro/IDO | Phase 2: CRS-207/Pembro
All-Cause Mortality (participants affected / at risk) | 8/8 | 3/4 | 7/16 | 1/1 | 1/3
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/4 | 9/16 | 1/1 | 1/3
Other Adverse Events (participants affected / at risk) | 8/8 | 4/4 | 16/16 | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: CRS-207 (N=8) | Phase 1: CRS-207/IDO 100 mg (N=4) | Phase 1: CRS-207/IDO 300 mg (N=16) | Phase 2: CRS-207/Pembro/IDO (N=1) | Phase 2: CRS-207/Pembro (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: CRS-207 (N=8) | Phase 1: CRS-207/IDO 100 mg (N=4) | Phase 1: CRS-207/IDO 300 mg (N=16) | Phase 2: CRS-207/Pembro/IDO (N=1) | Phase 2: CRS-207/Pembro (N=3)
Nausea (Gastrointestinal disorders) | 6 | 1 | 10 | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 1 | 9 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 8 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 6 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 4 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 4 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Lip blister (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 7 | 4 | 12 | 1 | 3
Pyrexia (General disorders) | 7 | 2 | 14 | 0 | 2
Fatigue (General disorders) | 3 | 2 | 11 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 3 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 2 | 0 | 0
Malaise (General disorders) | 1 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 2 | 0 | 0
Pain (General disorders) | 1 | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0
Hunger (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 2 | 10 | 0 | 2
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 5 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 5 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 6 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 2 | 5 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 5 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 4 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 3 | 2 | 3 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Listeriosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Bruxism (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 2 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
Study was terminated early and included a small number of subjects, and insufficient data were available to evaluate the clinical activity of the study treatment. Due to low enrollment, some protocol-specified outcome measures were not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction is that study results will first be published in a joint multi-center paper unless (a) written confirmation is provided to the site or PI indicating that there will be no multi-center publication, or (b) at least 12 months have passed after the completion of data analysis at all study sites. Publications will be submitted for sponsor review ≥ 45 days prior to the publication date. Sponsor cannot require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-02-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT02575807/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT02575807/SAP_001.pdf